CLINICAL TRIAL: NCT01546272
Title: Medico-economic Evaluation of Subcutaneous Automatic Resorbable Staples Device
Acronym: S2CARA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RC11_0147
Record Dates: First submitted 2012-02-21; First posted 2012-03-07 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: ENT Surgery; Gynecological Surgery; Plastic Surgery
Keywords: Subcutaneous resorbable sutures; Tolerance / effectiveness of subcutaneous suture; Reduced operative time and anesthesia time; Medico-economic evaluation; Accidental exposure to blood

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resorbable staples (Experimental): Suture using Insorb Resorbable staples
  Interventions: Device: Insorb resorbable staples
- Resorbable wires (Active Comparator): Suture using Monocryl resorbable wire
  Interventions: Device: Monocryl resorbable wire

INTERVENTIONS:
Device: Insorb resorbable staples — Subcutanous suture using resorbable staples
  Other Names: Insorb staples
  Arms: Resorbable staples
Device: Monocryl resorbable wire — Subcutanous suture using resorbable wire
  Other Names: Monocryl Wire
  Arms: Resorbable wires

SUMMARY:
A surgery made by an external incision requires to stitch the subcutaneous plans, usually performed using absorbable synthetic sutures hold on wire needle. This national, prospective, multicentric, and randomized study is devoted to estimate a technique of suture of the subcutaneous plans based on an implantable medical device delivering automatically absorbable staples. This particularly innovative technique lets to expect a tolerance and an efficiency at least equivalent to the reference technique (main objective). Moreover, this technique allows to anticipate a reduction of the duration of surgical procedure and anesthetic time while limiting the risks of blood wounds of the medical staff.The medical economic part of this study will check, from the point of view of the health care hospital, wether the technique is likely to reduce the costs and time consuming theater room procedures.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 yrs to 75 yrs
* Patient supported for a scheduled surgery :

For abdominoplasty, cervicotomy or suprapubic surgery With a open incision necessary for operative exposition of 10 cm or more with a straight or curved surgery incision

* Person covered by Health Insurance
* ECOG Performance Status 0 or 1
* Patient's informed and written consent

Exclusion Criteria:

* Incision imposing a very angular or sinuous scar for which the use of the medical device is deemed unsuited (sinuous or bayonet incisions)
* Known history of intolerance to any component of the medical device
* Immunocompromised patients or undergoing a long term treatment by corticosteroids or immunosuppressants
* Known or anticipated presence of a skin infection (due to the infected skin condition, or because of underlying surgery conducted in infected territory or likely to be)
* Dermatological disease or skin treatment in progress
* History of radiation therapy on the surgical site or antimitotic treatment in progress
* Pregnancy at the time of suture
* Patients simultaneously included in another treatment protocol
* Patients under legal guardianship
* Non French speaking patients, refusing or unfit for the monitoring proposed in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 664 (Actual)
Dates: Start 2012-03; Primary Completion 2014-05 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Overall PSAS score measured 3 months after the surgery | 3 months after the surgery
  Overall PSAS score measured 3 months after the surgery(PSAS : "Patient Scar Assessment Scale")

SECONDARY OUTCOMES:
Incremental cost-effectiveness ratio (ICER) or average cost of suture according to the procedure (wire or staple) | Day 0 (Procedure)
Presence of scarring complications at day 8 (infection, dehiscence) | Day 8
Measurement of suture, surgical and anesthetic times | Day 0 (procedure)
Overall score of the PSAS scale | Months 3, 12 and 18
  The tolerance will be assessed by the overall score of the PSAS scale (Patient Scar Assessment Scale)
Overall score of the OSAS scale | Months 3, 12 and 18
  The scar quality will be assessed by the overall score of the OSAS scale (Observer Scar Assessment Scale)
Aesthetic quality of the scar | Month 18
  The aesthetic quality of the scar will be assessed by the patient and a physician (not the surgeon) by a score range from 0 to 10
Quantification of accidental exposure to blood | During the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Malard, Professor, Principal Investigator — Nantes University Hospital
Locations (24):
- France (24):
  - CHU de Nantes, Nantes, Pays de la Loire Region
  - Amiens University Hospital, Amiens
  - Angers University Hospital, Angers
  - Besançon University Hospital, Besançon
  - Bordeaux University Hospital "Centre FX. Michelet", Bordeaux
  - Brest University Hospital "Hôpital du Morvan", Brest
  - Caen University Hospital "Hôpital de la Côte de Nacre", Caen
  - Lille University Hospital "Hôpital Roger Salengro", Lille
  - "Assistance Publique des Hôpitaux de Marseille - La Conception", Marseille
  - Montpellier University Hospital "Hôpital Gui de Chauliac", Montpellier
  - Mulhouse Hospital "Emile Muller", Mulhouse
  - CHU Nantes, Nantes
  - "Institut de Cancérologie de Nice", Nice
  - "Assistance Publique des Hôpitaux de Paris - Hôpital Bichat", Paris
  - CHU Poitiers, Poitiers
  - Poitiers University Hospital, Poitiers
  - Rennes University Hospital "CHU Pontchaillou", Rennes
  - Rennes University Hospital, Rennes
  - Rouen University Hospital, Rouen
  - Strasbourg University Hospital "Hôpital Hautepierre", Strasbourg
  - "Institut Claudius Regaud", Toulouse
  - "Pôle Santé Léonard de Vinci", Tours
  - Pôle Santé Léonard de Vinci, Tours
  - Tours University Hospital, Tours